CLINICAL TRIAL: NCT03270917
Title: The ORANGE SEGMENTS - Trial: an International Multicentre Randomized Controlled Trial of Open Versus Laparoscopic Parenchymal Preserving Postero-superior Liver Segment Resection
Brief Title: ORANGE SEGMENTS: Open Versus Laparoscopic Parenchymal Preserving Postero-Superior Liver Segment Resection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); The Queen Elizabeth Hospital (Other); General Hospital Groeninge (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); King's College Hospital NHS Trust (Other); San Raffaele University Hospital, Italy (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Oslo University Hospital (Other); Oxford University Hospitals NHS Trust (Other); Derriford Hospital (Other); University Hospital Southampton NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Moscow Clinical Scientific Center (Other); San Camillo Hospital, Rome (Other); Fondazione Poliambulanza Istituto Ospedaliero (Other); Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL36215.068.11*
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Liver Surgery
Keywords: Parenchymal preserving; Postero-superior; Laparoscopy; Hepatectomy

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to either the open or the laparoscopic treatment arm.
Who Masked: Participant, Investigator
Masking Description: The patient, ward physician and research investigator are blinded to the treatment intervention. A large abdominal dressing will be used to cover the incision(s) until postoperative day 4. Obviously, the surgeon and anaesthesiology team can not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open (Other): Open liver surgery
  Interventions: Procedure: Parenchymal preserving postero-superior liver segment resection
- Laparoscopy (Other): Laparoscopic liver surgery
  Interventions: Procedure: Parenchymal preserving postero-superior liver segment resection

INTERVENTIONS:
Procedure: Parenchymal preserving postero-superior liver segment resection — Parenchymal preserving liver segment resection of one or two of the postero-superior liver segments (4A, 7 or 8).

SUMMARY:
The international and multicentre ORANGE SEGMENTS - Trial is a prospective, double blinded, randomized controlled study comparing patients undergoing parenchymal preserving resection of postero-superior liver segments (involving one or two of segments 4a, 7, 8). All patients will be participating in an enhanced recovery programme.

Primary outcome is time to functional recovery. Secondary study parameters include hospital length of stay, intraoperative blood loss, operation time, liver specific morbidity, readmission percentage, resection margin, quality of life, body image and cosmesis , reasons for delay of discharge after functional recovery, long term incidence of incisional hernias, hospital and societal costs during one year, time to adjuvant chemotherapy initiation, overall five-year survival.

DETAILED DESCRIPTION:
Liver resection for colorectal metastasis is a potential curative therapy and has become the standard of care in appropriately staged patients, offering five-year survival rates ranging from 38 up to 61% in selected cases, with approximately 30% of patients surviving ten years or more, compared to five-year survival rates of less than 5% for patients not amenable to resection. Liver surgery is also a widely accepted treatment for symptomatic benign lesions and those of uncertain nature or large size. Whilst the figures are a vast improvement on the past, there is still a need to refine the treatment of these patients, including surgical technique.

Open hepatectomy is the current standard of care for the management of primary and secondary tumours. The open postero-superior liver segment resection requires a large incision to achieve adequate access and proper control during resection. This has a significant impact on patient's recovery and, in cases of small resections, this access may represent the major component of surgical trauma. Advances in surgical technique and expertise now permit these operations to be performed with minor incisions by using the laparoscopic approach. Although the feasibility of laparoscopic hepatectomy has been established, only select centres use this technique as their primary modality.

Laparoscopic liver resection was first reported in 1991. Over the past decades, the method has gained wide acceptance for various liver resection procedures. Multiple retrospective case series, patient cohorts, systematic reviews and meta-analyses have compared open with laparoscopic liver surgery and indicate the laparoscopic approach to be safely applicable for the resection of both malignant and benign liver lesions. Laparoscopic liver resection has been associated with shorter hospital length of stay, reduced intraoperative blood loss, less postoperative pain and earlier recovery. Despite this, concerns remain over operative times, the ability to control haemorrhage laparascopically and long-term oncological outcomes.

Initially, the left lateral segments of the liver were chosen for anatomic laparoscopic resection, with good results. Many liver centres worldwide currently use laparoscopy for resection of the anterior liver segments. Whilst case control studies would now seem sufficient to allay such concerns in the context of minor liver resections and left lateral sectionectomies, the adoption and dissemination of laparoscopy by hepatobiliary oncologic surgeons for major hepatectomies and resections of postero-superior segments has been restricted. Besides the relatively low volume of patients, major laparoscopic liver resections are technically demanding, have a significant learning curve, are time consuming, are thought to hold an increased morbidity risk and lack in evidence.

Nevertheless, a new impulse for the laparoscopic management of major liver lesions came after the first reports of laparoscopic hemihepatectomies, which demonstrated that in expert hands major anatomical laparoscopic liver resections are feasible with good efficacy and safety. When comparing surgical procedures, one of the easiest to measure and often used outcomes is the length of hospital stay; the time it takes for a patient to be discharged from the hospital after an operation. On the whole, a median hospital length of stay of 6.0 to 13.1 days and 3.5 to 10.0 days have been observed after open and laparoscopic hepatic resections in European centres respectively. For major surgery in expert centres, median duration of hospital admission varied between 6 to 12.5 days for open surgery and 4 to 8.2 days for laparoscopic resections. Concentrating on postero-superior liver segment resections, the median hospital stay is 6 days (3-44 days) for those undergoing open compared with 4 days (1-11 days) for those having laparoscopic resections.

Besides the immediate benefits to the patient, such as decreased intraoperative blood loss, diminished postoperative pain, earlier recovery and reduced hospital length of stay, laparoscopic liver surgery may also have the potential to improve outcomes in the longer term by reducing complications, enhancing quality of life, improving cosmesis, ensuring early commencement and completion of adjuvant therapies. However, level-1 evidence on all outcomes is still to be presented.

Within the framework of optimized perioperative care, broader indications for hepatic surgery and further adoption of laparoscopic liver resections, there is a clear need for a randomized trial. Therefore, the multicentre and international ORANGE SEGMENTS - Trial has been designed to provide evidence on the merits of laparoscopic versus open parenchymal preserving postero-superior liver segment resection within an enhanced recovery programme in terms of time to functional recovery, hospital length of stay, intraoperative blood loss, operation time, resection margin, time to adjuvant chemotherapy initiation, readmission percentage, (liver specific) morbidity, quality of life, body image, reasons for delay of discharge after functional recovery, long term incidence of incisional hernias, hospital and societal costs during one year and overall five-year survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a parenchymal sparing liver resection (including wedge resections and full segmentectomies) involving one or two of segments 4a/7/8 for accepted indications . A segment 6/7 resection would also be eligible.
* Able to understand the nature of the study and what will be required of them.
* Men and non-pregnant, non-lactating women, aged 18 years and older.
* BMI between and including 18-35 kg/m2
* Patients with ASA physical status I-II-III.

Exclusion Criteria:

* Inability to give (written) informed consent.
* Patients requiring other liver surgery than a parenchymal sparing resection involving one or two of segments 4a, 7, 8.
* Patients requiring parenchymal sparing liver resection involving segment 1. This is due to the high level of technical difficulty.
* Patients with hepatic lesion(s), that are located with insufficient margin from vascular or biliary structures to be operated laparoscopically.
* Patients with ASA physical status IV-V.
* Repeat hepatectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to functional recovery | expected average of 4-10 days
  Time until a patient is functionally recovered

SECONDARY OUTCOMES:
Hospital length of stay | 30 days
  Total length of hospital stay
Intraoperative blood loss | during procedure
  Net intraoperative blood loss
Operating time | surgical time from incision until closure
(Liver specific) morbidity | 1 year
  Composite endpoint of liver specific morbidity (intra-abdominal bleeding, intra-abdominal abcess, ascites, postresectional liver failure, intra-operative mortality, bile leakage)
Readmission percentage | 1 year
  Total percentage of patients being readmitted
Resection margin | 1 year
  Residual tumor cells in resection border
Quality of life | 1 year
  The physical, social and emotional well-being of the patient
Body image and cosmesis | 1 year
  The aesthetic appearance of the scars associated with the operation and its influence on the patient self-view
Reasons for delay of discharge after functional recovery | 1 year
  All reasons that may cause delay in discharge after the patient has recovered functionally, such as administrative reasons, patient confidence, logistics problems, etc.
Incisional herniation | 1 year
  Cicatricial hernia
Hospital and societal costs | 1 year
  All costs that are associated with the operation, including in-hospital costs and out of hospital costs, such as home care, work absence, etc.
Time to adjuvant chemotherapy initiation | 1 year
  The time it takes to start adjuvant chemotherapy after the patient has been operated
Overall five-year survival | 5 years
  Five-year survival

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abu Hilal, Prof., Study Chair — University Hospital Southampton NHS Foundation Trust; John Primrose, Prof., Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (16):
- General Hospital Groeninge, Kortrijk, Belgium
- Italy (3):
  - Poliambulanza Hospital, Brescia
  - San Raffaele Hospital, Milan
  - San Camillo-Forlanini Hospital, Rome
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Maastricht University Medical Center+, Maastricht
- University Hospital Oslo, Oslo, Norway
- Moscow Clinical Scientific Center, Moscow, Russia
- United Kingdom (8):
  - Aintree University Hospital, Aintree
  - Queen Elizabeth Hospital, Birmingham
  - King's College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle
  - Oxford University Hospitals, Oxford
  - Derriford Hospital, Plymouth
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coles SR, Besselink MG, Serin KR, Alsaati H, Di Gioia P, Samim M, Pearce NW, Abu Hilal M. Total laparoscopic management of lesions involving liver segment 7. Surg Endosc. 2015 Nov;29(11):3190-5. doi: 10.1007/s00464-014-4052-2. Epub 2015 Jan 13. PMID 25582963
- [Background] Cipriani F, Shelat VG, Rawashdeh M, Francone E, Aldrighetti L, Takhar A, Armstrong T, Pearce NW, Abu Hilal M. Laparoscopic Parenchymal-Sparing Resections for Nonperipheral Liver Lesions, the Diamond Technique: Technical Aspects, Clinical Outcomes, and Oncologic Efficiency. J Am Coll Surg. 2015 Aug;221(2):265-72. doi: 10.1016/j.jamcollsurg.2015.03.029. Epub 2015 Mar 27. PMID 25899733
- [Background] Scuderi V, Barkhatov L, Montalti R, Ratti F, Cipriani F, Pardo F, Tranchart H, Dagher I, Rotellar F, Abu Hilal M, Edwin B, Vivarelli M, Aldrighetti L, Troisi RI. Outcome after laparoscopic and open resections of posterosuperior segments of the liver. Br J Surg. 2017 May;104(6):751-759. doi: 10.1002/bjs.10489. Epub 2017 Feb 13. PMID 28194774
- [Background] Zheng B, Zhao R, Li X, Li B. Comparison of laparoscopic liver resection for lesions located in anterolateral and posterosuperior segments: a meta-analysis. Surg Endosc. 2017 Nov;31(11):4641-4648. doi: 10.1007/s00464-017-5527-8. Epub 2017 Apr 7. PMID 28389796
- [Derived] Sijberden JP, Kuemmerli C, Ratti F, D'Hondt M, Sutcliffe RP, Troisi RI, Efanov M, Fichtinger RS, Diaz-Nieto R, Ettorre GM, Sheen AJ, Menon KV, Besselink MG, Soonawalla Z, Aroori S, Marino R, De Meyere C, Marudanayagam R, Zimmitti G, Olij B, Eminton Z, Brandts L, Ferrari C, M van Dam R, Aldrighetti LA, Pugh S, Primrose JN, Abu Hilal M. Laparoscopic versus open parenchymal preserving liver resections in the posterosuperior segments (ORANGE Segments): a multicentre, single-blind, randomised controlled trial. Lancet Reg Health Eur. 2025 Feb 20;51:101228. doi: 10.1016/j.lanepe.2025.101228. eCollection 2025 Apr. PMID 40060302
- [Derived] Kuemmerli C, Fichtinger RS, Moekotte A, Aldrighetti LA, Aroori S, Besselink MGH, D'Hondt M, Diaz-Nieto R, Edwin B, Efanov M, Ettorre GM, Menon KV, Sheen AJ, Soonawalla Z, Sutcliffe R, Troisi RI, White SA, Brandts L, van Breukelen GJP, Sijberden J, Pugh SA, Eminton Z, Primrose JN, van Dam R, Hilal MA; ORANGE trials collaborative. Laparoscopic versus open resections in the posterosuperior liver segments within an enhanced recovery programme (ORANGE Segments): study protocol for a multicentre randomised controlled trial. Trials. 2022 Mar 9;23(1):206. doi: 10.1186/s13063-022-06112-3. PMID 35264216